CLINICAL TRIAL: NCT05026567
Title: A Single Center, Single Dose, Open Label, Randomized, Four-period Crossover Study in Healthy Subjects to Describe and Compare the Plasma Pharmacokinetics of Midazolam After Intramuscular Injection as a Solution by a Conventional Syringe or by the Needle-free Injector ZENEO®
Brief Title: Bioavailability Study of Midazolam Administered as a Solution by Conventional Syringe or ZENEO®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crossject (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJTPKL172001
Record Dates: First submitted 2021-07-19; First posted 2021-08-30 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reference Product A (Active Comparator)
  Interventions: Drug: 2 ml of DORMICUM® Midazolam Hydrochloride (15 mg/3 mL)
- Experimental B (Experimental)
  Interventions: Combination Product: ZENEO® Midazolam (10 mg/0.625 mL) on bare skin in thigh
- Experimental C (Experimental)
  Interventions: Combination Product: ZENEO® Midazolam (10 mg / 0.625 mL) on bare skin in ventrogluteal area
- Experiment D (Experimental)
  Interventions: Combination Product: ZENEO® Midazolam (10 mg / 0.625 mL) through clothing in thigh

INTERVENTIONS:
Drug: 2 ml of DORMICUM® Midazolam Hydrochloride (15 mg/3 mL) — Intramuscular injection
  Arms: Reference Product A
Combination Product: ZENEO® Midazolam (10 mg/0.625 mL) on bare skin in thigh — Intramuscular injection
  Arms: Experimental B
Combination Product: ZENEO® Midazolam (10 mg / 0.625 mL) on bare skin in ventrogluteal area — Intramuscular injection
  Arms: Experimental C
Combination Product: ZENEO® Midazolam (10 mg / 0.625 mL) through clothing in thigh — Intramuscular injection
  Arms: Experiment D

SUMMARY:
Primary objective of this study is to describe the plasma pharmacokinetics of midazolam after single intramuscular injection on bare skin in the thigh by the needle-free injector Zeneo® compared to injection on bare skin in the thigh by a conventional syringe (Reference) in terms of relative bioavailability and bioequivalence.

DETAILED DESCRIPTION:
Secondary objectives are:

* To describe the plasma pharmacokinetics of midazolam after single intramuscular injection on bare skin in the ventrogluteal area by the needle-free injector Zeneo® compared to injection on bare skin in the thigh by a conventional syringe (Reference) in terms of relative bioavailability and bioequivalence.
* To describe the plasma pharmacokinetics of midazolam after single intramuscular injection through clothing in the thigh by the needle-free injector Zeneo® compared to injection on bare skin in the thigh by a conventional syringe (Reference) in terms of relative bioavailability and bioequivalence.
* To describe the plasma pharmacokinetics of midazolam after single intramuscular injection through clothing in the thigh by the needle-free injector Zeneo® compared to injection on bare skin in the thigh by the needle-free injector Zeneo® in terms of relative bioavailability and bioequivalence.
* To describe the plasma pharmacokinetics of midazolam after single intramuscular injection on bare skin in the thigh by the needle-free injector Zeneo® compared to injection on bare skin in the ventrogluteal area by the needle-free injector Zeneo® in terms of relative bioavailability and bioequivalence
* To assess and compare the pharmacokinetics of the major active metabolite 1'-OH midazolam after a single intramuscular injection i.m. administration when delivered by ZENEO®® orvs. administration by conventional syringe (Reference)conventional syringe with needle.
* To assess and compare the pharmacokinetics of ZENEO® Midazolam (10mg / 0.625mL) administered in the thigh on bare skin and ZENEO® Midazolam (10mg / 0.625mL) administered in the thigh through clothing.
* To assess safety and tolerability of midazolam after a single intramuscular injection single i.m. administration whenby delivered by ZENEO® vs. administrationor by conventional syringe (Reference) by conventional syringe with needle.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, 18 to 59 years (inclusive) at screening.
2. Body Mass Index (BMI) between 18.5 and 29.9 kg/m2 (inclusive).
3. Body mass weight between 50 and 110 kg (inclusive)
4. Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
5. Non-smokers or past-smokers who stopped at least 3 months before the study.
6. Female subject must be either of

   * non-childbearing potential: post-menopausal (defined as at least 1 year without any menses) prior to Screening, or documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening).
   * or, if of childbearing potential, must have a negative serum pregnancy test at Screening and must use two forms of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 28 days [or 5 half-lives of the study drug whichever is longer] after the final study drug administration. Acceptable forms of birth control include: placement of a non-hormonal intrauterine device or intrauterine system, 2) barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) or abstinence of male/female intercourse if it is a part of normal practice in her life.

   The use of hormonal contraception in this study is not allowed. For male subjects contraception is not needed during this study.
7. Injection sites must be clear of tattoos, scars and moles.
8. Signed written consent given for participation in the study.

Exclusion Criteria:

1. Any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease, as judged by the Investigator.
2. Medical history of malignant disease (with the exception of localized skin or cervical carcinoma that had been excised and cured)
3. Any clinically significant abnormality following the Investigator's review of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or admission to the clinical unit.
4. A pulse < 40 or > 100 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (measurements taken in triplicate after subject has been resting in supine position for 5 minutes.
5. A mean corrected QT interval using Fridericia's formula (QTcF) interval > 450 ms at screening. If the mean QTcF exceeds the limits above, one additional triplicate ECG may be taken. If this triplicate also gives an abnormal result, the subject should be excluded.
6. History of smoking within 3 months prior to the first admission to the clinical unit.
7. History of drinking more than 21 units of alcohol per week (1 unit = 10 g pure alcohol = 250 ml of beer [5%] or 35 ml of spirits [35%] or 100 ml of wine [12%]) within 3 months prior to the first admission to the clinical unit.
8. Any recreational use of drugs-of-abuse within 3 months prior to the first administration of an IMP.
9. Use of any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to first study medication administration, except for the occasional use of paracetamol (up to 2 g/day)- except if it will not affect the study outcome at the discretion of the investigator.
10. Use of drugs that induce hepatic enzymes (rifampicin, rifabutin, carbamazepine, phenobarbitone, phenytoin, primidone, and aminoglutethimide).
11. Use of inhibitors of the CYP3A4 enzyme (including but not only clarithromycin, itraconazole, erythromycin, fluconazole, verapamil). (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)
12. Participation in any clinical study within 3 months prior to the expected date of enrolment into the clinical study, provided that the clinical study did not entail a biological compound with a long half-life or participation in more than 3 clinical studies within 12 months.
13. Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
14. A major illness during the 3 months before commencement of the screening period.
15. Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
16. Any significant blood loss, donated one unit (450 m) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to the first admission to the clinical unit.
17. History of hypersensitivity or allergy to the IMP or its excipients or any related medication.
18. The subject has any other condition, which in the opinion of the Investigator precludes the subject's participation in the clinical study, including any conditions mentioned in contraindication, special warnings and precautions for use, in the summary of product characteristics of the IMP.
19. History of COVID illness in last 30 days.
20. Positive serology test for hepatitis B surface antigen, hepatitis C virus antibodies or human immunodeficiency virus-1 and/or 2 antibodies.
21. Positive pregnancy test.
22. Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
23. Positive urine screen for tobacco use.
24. Any specific investigational product safety concern.
25. Vulnerable subjects, e.g. persons in detention.
26. Employee of the sponsor (or authorized representative), or FARMOVS (or authorized representative)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve, time zero to time of the last quantifiable concentration (AUC0-t) | up to 36hours
Area under the plasma concentration versus time curve, with extrapolation to infinity (AUC0-∞) | up to 36hours
Maximum observed plasma concentration Cmax | up to 36hours

SECONDARY OUTCOMES:
Time to peak drug concentration (Tmax) of midazolam | up to 36 hours
Terminal half-life (T1/2) of midazolam | up to 36 hours
Time to peak drug concentration (Tmax) of 1'OH-midazolam | up to 36 hours
Terminal half-life (T1/2) of 1'OH-midazolam | up to 36 hours
Maximum observed plasma concentration (Cmax) 1'OH-midazolam | up to 36 hours
Area under the plasma concentration versus time curve from time 0 to the last measurable concentration (AUC0-t) of 1'OH-midazolam | up to 36 hours
Area under the plasma concentration versus time curve from time 0 extrapolated to infinite time (AUC0- ∞) of 1'OH-midazolam | up to 36 hours
Pain evaluation using the visual analogue scale (0:no pain-10:pain as bad as it could possibly be) | up to 5 hours
Number of Safety/adverse events | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: EFW Krantz, PhD, Principal Investigator — Farmovs
Locations (1):
- FARMOVS Pty Ltd, Bloemfontein, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacombe O, Pletan Y, Grouin JM, Brennan A, Gire O. Relative Bioavailability Study of Midazolam Intramuscularly Administered with the Needle-Free Auto-Injector ZENEO(R) in Healthy Adults. Neurol Ther. 2024 Aug;13(4):1155-1172. doi: 10.1007/s40120-024-00627-4. Epub 2024 May 28. PMID 38806873